CLINICAL TRIAL: NCT04856605
Title: The Factors Associated With Occurrence and Healing Of Umbilical Pilonidal Sinus Disease
Brief Title: Umblical Pilonidal Sinus Evaluation
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Arda Isik, MD, FEBS, FACS, assoc.prof., Istanbul Medeniyet University
Other Study IDs: umblicalps
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — regular surgery

SUMMARY:
Purpose: Pilonidal sinus disease (PSD) is a chronic inflammatory condition of skin due to implanted loose hair. PSD is commonly seen in sacrococcygeal region, but can also be seen in axilla, perineum, suprapubic regions, on hands and umbilicus. The aim of this project was to find factors influencing the development and treatment of umbilical pilonidal sinus.

Material and methods: In this cross-sectional prospective study, the investigators evaulated 82 (19 female, 63 male) patients with a history of umbilical pilonidal disease (e.g. predisposing factors, treatment modalities) between 2012 and 2020.

DETAILED DESCRIPTION:
In this study, participants were volunteer patients admitted to Erzincan University Medical Faculty to the General Surgery Outpatient Clinic between March of 2012 and December of 2020 with umbilical symptoms such as umbilical discharge and umbilical pain. All patients were diagnosed by physical examination confirmed with ultrasonography . Patients with diseases other than umbilical sinus were excluded from the study. Examined patients' characteristics include age, gender, intergluteal sinus disease history, family history, belly shaving histoy, daily shower, treatment modality and healing status. There were 3 treatment modalities: conservative approach (daily shower, shaving, antibitics if infected); topical silver nitrate treatment; surgical operation for umbilical sinus as excracting the hairs from the sinus ± excising the sinus. To determine if "healed" the investigators followed up our patients ensuring no symptoms for a minimum 2 years.

Chi-square tests were conducted to compare the distribution of categorical variables. Age was analyzed as a continuous variable with a t-test. Univariable and multivariable logistic regression models were used to calculate odds ratios and 95% confidence intervals. P-values of less than 0.05 were considered statistically significant. Statistical analyses were conducted with R version of 3.6.1 (R Foundation for Statistical Computing, Vienna, Austria, https://www.r-project.org) software packages.

ELIGIBILITY:
Inclusion Criteria:

* all patients with umblical pilonidal sinus

Exclusion Criteria:

* no disease

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients who have umblical pilonidal disease
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
healing status | 2 year
  to define the best method for healing. It will be measured by the duration(days) of healing.

SECONDARY OUTCOMES:
recurrence status | 2 year
  to define the best method for recurrence prevention. Recurrence will be noted as purulent discharge over the umblicus.

OTHER OUTCOMES:
duration of wound healing | 2 year
  The investigators will measure the diameter(cm) of the wound everyday.

CONTACTS AND LOCATIONS:
Overall Officials: ARDA ISIK, Principal Investigator — MEDENIYET UNIVERSITY

IPD SHARING:
Plan to Share IPD: No